CLINICAL TRIAL: NCT05825846
Title: Impact of Slow Breathing on Markers of Stress in Response to a Virtual Reality Active Shooter Drill
Brief Title: Impact of Breathing Interventions on Stress Markers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Texas State University (Other)
Collaborators: M. Hunter Martaindale (Unknown); C. Dillard (Unknown); S. Hunter (Unknown)
Responsible Party: Principal Investigator, Matt McAllister, Associate Professor, Texas State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Breathing and VR-ASD
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Physiological Stress

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to one of two treatments:
  1. slow breathing 1 (SB1)
  2. slow breathing 2 (SB2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow breathing 1 (SB1) (Experimental): Four second inhale through the nasal + hold two seconds + four second exhale through the mouth + hold for two seconds, repeat (~25 breath cycles within the 5 min intervention)
  Interventions: Device: Virtual- reality active shooter drill
- Slow breathing 2 (SB2) (Experimental): Four second inhale through the nose into the diaphragm followed by a two second exhale, repeat (~50 breath cycles within the 5 min intervention)
  Interventions: Device: Virtual- reality active shooter drill

INTERVENTIONS:
Device: Virtual- reality active shooter drill — The stress protocol used for this experiment utilized a previously studied virtual reality active shooter drill (VR-ASD). The VR-ASD scenario (~2 min) involves the participant physically walking down a ~10-foot-long virtual hallway where they will encounter wounded victims. Once at the threshold of to the attack room, they will observe one victim on the ground with a traumatic head injury and the shooter firing his handgun at the last victim, the participant will "fire" a shot, and the shooter will fall after being shot.

SUMMARY:
The goal of this clinical trial is to examine the effects of slow breathing breathing on markers of stress in healthy college aged individuals. The breathing intervention is performed for five minutes pre and post a virtual reality active shooter drill.

The main question to answer is:

1) what is the impact of a controlled breathing intervention and virtual reality active shooter drill on markers of subjective and biological stress?

DETAILED DESCRIPTION:
For this study participants will be randomly assigned either slow breathing 1 [(SB1); four second inhale, two second pause, four second exhale, two second pause, repeat for five minutes] or slow breathing 2 [(SB2); four second inhale, two second exhale, repeat for five minutes]. The breathing intervention will take place five minutes prior to the start of the virtual reality based active shooter drill. Researchers will compare the two groups in terms of change in heart rate (HR), blood pressure (BP) subjective stress [(SAI); state-trait anxiety inventory], and salivary markers of stress before and after the breathing intervention and virtual reality active shooter drill (VR-ASD).

All procedures were reviewed and approved by the University Institutional Review Board.

Experimental procedures upon arrival to the testing site, subjects will be instructed to rinse their mouth with water and rest in a quiet room for 10 minutes. Immediately after the 10 minutes of rest period, an initial saliva sample, HR & BP (Suntech, Hauppauge, NY, USA) and SAI measures were collected (30 min prior to VR-ASD). Throughout the experimental session HR, BP, SAI, and saliva samples will be collected a total of four times : 1) 30 minutes prior to start of the VR-ASD, 2) 5 minutes prior to the start of the VR-ASD (immediately before the breathing intervention) 3) 5 minutes post VR-ASD (immediately post breathing intervention), and 4) 30 minutes post VR-ASD.

Virtual Reality- Active Shooter Drill (VR-ASD):

This is a virtually reality simulation, the participant will put on the VR headset and carry a Glock 17 training pistol, they will be able to physically move through the entire ASD without interruption. The VR lab is larger than the virtual environment (~35 x 20 ft). The participant will physically walk down a ~10-foot-long virtual hallway where they will encounter 2 simulated wounded victims. One will be on the ground with traumatic injuries and the second victim will 'run' out of the attack room with gunshot wounds to his/her left arm and leg. Once at the threshold of to the attack room, they will observe one victim on the ground with a traumatic head injury and the shooter firing his handgun at the last victim. If the subject hadn't fired his/her weapon yet, the shooter would turn toward the participant to elicit a response, the participant will " fire" a shot if needed. The shooter will fall after being shot.

Slow breathing 1 ("Box" breathing/slow breathing): Four second inhale through the nasal + hold two seconds + four second exhale through the mouth + hold for two seconds, repeat (~25 breath cycles within the 5 min intervention) Slow breathing 2: Four second inhale through the nose into the diaphragm followed by a two second exhale, repeat (~50 breath cycles within the 5 min intervention)

Breathing Instructional video The lead researcher will provide a 5- minute instructional video over randomly assigned breathing method to the participant prior to starting the breathing intervention. The instructional video will include a visual of the researcher performing the breathing intervention alongside a voice over with a countdown on the screen to go-along with the breathing tempo. A researcher will be in the room with the participant counting their breaths per minute to make sure they are keeping up with the breathing tempo and ending at the appropriate time. If the participant is unable to keep up with the breathing tempo they will be asked to discontinue.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy, aged 18-39
* free from any known cardiovascular or metabolic diseases,
* free from any major stressors within the last 30 days such as birth of a child, abortion, or divorce.

Exclusion Criteria:

* subjects are required to not have a history of motion sickness, or vertigo
* not previously diagnosed with a brain injury or epilepsy, asthma, or currently taking psychological medication

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
salivary secretory IgA | Up to 8 months
  SIgA is a marker of immune function and salivary SIgA concentrations tend to increase when exposed to stress
salivary alpha amylase | up to 8months
  salivary alpha amylase is an enzyme involved in digestive processes. Amylase concentration in saliva have been shown to reflect sympathetic stress. Thus, as sympathetic stress increases, salivary amylase concentrations tend to increase.
salivary cortisol | up to 8 months
  salivary cortisol is a marker of stress which reflects activation on the hypothalamic pituitary adrenal axis
heart rate | Up to 8 months
  heart rate reflects activity from parasympathetic and sympathetic nervous system and increases when exposed to stress
State trait anxiety inventory | Up to 8 months
  state anxiety inventory is a subjective scale which includes six short statements such as "I feel calm" or "I feel tense" and composite scores of participant responses are used for analysis. Higher values reflect higher subjected anxiety.
systolic and diastolic blood pressure | Up to 8 months
  Blood pressure measures the force and pressure of blood in the arteries. When stressed the activation of the autonomic nervous system produces vasoconstricting hormones and releases them when exposed to stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas State University, San Marcos, Texas, United States

REFERENCES:
- [Derived] Dillard CC, Martaindale H, Hunter SD, McAllister MJ. Slow Breathing Reduces Biomarkers of Stress in Response to a Virtual Reality Active Shooter Training Drill. Healthcare (Basel). 2023 Aug 21;11(16):2351. doi: 10.3390/healthcare11162351. PMID 37628548